CLINICAL TRIAL: NCT07267442
Title: Turkish Translation , Validity and Reliability of the Hypertonia Assessment Tool in Children With Motor Disorders
Status: Recruiting | Type: Observational
Sponsor: Kastamonu University (Other)
Collaborators: Gazi University (Other)
Responsible Party: Principal Investigator, Hidayet Cuha, Lecturer, PT, PhD(c), Kastamonu University
Other Study IDs: 2024 - 1944
Record Dates: First submitted 2025-11-23; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Motor Disorder; Reliability and Validity; Hypertonia
Keywords: Hypertonia; Motor Disorder; Reliability and Validity
MeSH Terms: conditions — Motor Disorders; Muscle Hypertonia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with motor disorders

SUMMARY:
Translating batteries with good psychometric properties into Turkish will increase the number of assessment batteries we can use in our language for clinical and academic studies. Therefore, the aim of our study was to verify the validity, reliability, and translation into Turkish of the Hypertonus Assessment Tool for children with motor disorders.

DETAILED DESCRIPTION:
Among children with omotor disorders, particularly those with cerebral palsy, abnormalities in muscle tone are among the most common clinical symptoms. Damage occurring in various structures such as the thalamus, cerebral cortex, and basal ganglia can adversely affect muscle tone. Hypertonia is defined as an abnormal increase in resistance to externally imposed movement about a joint. It leads to limitations in activity participation, loss of motor control, and reduced quality of life. Hypertonia, which causes impairments in gross motor skills such as walking, stair climbing, and crawling, negatively affects the quality of life in childhood.

Muscle tone disorders in childhood can be classified into three main types: spasticity, dystonia, and rigidity. Spasticity is defined as a velocity-dependent increase in muscle tone associated with hyperexcitability of the tonic stretch reflex. Dystonia is a movement disorder characterized by sustained or intermittent involuntary muscle contractions that cause twisting, repetitive movements, abnormal postures, or a combination of these. Rigidity refers to bidirectional, velocity-independent resistance to passive movement, which may involve simultaneous co-contraction of agonist and antagonist muscles. In some cases, more than one type of tone abnormality may coexist.

Several assessment tools have been developed to evaluate different subtypes of hypertonia or general increases in tone. The most commonly used methods in clinical and research settings include the Modified Ashworth Scale (MAS), the Modified Tardieu Scale (MTS), and the Barry-Albright Dystonia Scale (BADS). While these scales evaluate different aspects of hypertonia, they do not distinguish between its subtypes. The Hypertonia Assessment Tool (HAT) was developed to address the need for a single instrument capable of differentiating among hypertonia subtypes. Introduced to the literature by Fehlings et al. in 2010, the HAT has been shown to be a valid and reliable tool for assessing the three subtypes of hypertonia in children with cerebral palsy.

The HAT involves observing an extremity joint during passive stretch and voluntary movement to detect increased tone or resistance. The scale consists of seven items-two assessing spasticity, two rigidity, and three dystonia. It can differentiate hypertonia subtypes in both upper and lower extremities and takes approximately five minutes to administer per limb. Studies in various patient populations have reported moderate to good levels of validity and reliability.

Translating psychometrically robust assessment tools into Turkish will expand the number of instruments available for clinical and research use in our native language. Therefore, the aim of this study was to translate the Hypertonia Assessment Tool into Turkish and to evaluate its validity and reliability in children with motor disorders.

ELIGIBILITY:
Inclusion Criteria:

* as voluntary participation in the study,
* a diagnosis of a neuromotor disorder under the age of 18,
* sufficient cognitive ability to follow verbal commands

Exclusion Criteria:

* Patients with any other systemic disease,
* Who had received botulinum toxin A injections or undergone surgery within the past three months,
* Be unable to follow verbal instructions
* Medical treatment had been modified within the last month

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This methodological study was designed as a Turkish language adaptation, validity, and reliability study. It will be conducted at the Developmental Physiotherapy and Pediatric Rehabilitation Unit of the Department of Physiotherapy and Rehabilitation, Faculty of Health Sciences, Gazi University, between January 15, 2025, and January 15, 2026. Children with neuromotor disorders diagnosed by a pediatric neurologist and attending routine clinical follow-up visits will be recruited through convenience sampling. The total sample size was determined as 70 participants, corresponding to ten times the number of items in the scale. Children whose parents provide written and verbal informed consent will be included in the study.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2026-01-10 (Estimated); Study Completion 2026-06-10 (Estimated)

PRIMARY OUTCOMES:
Hypertonia Assessment Tool | The patient, diagnosed by a pediatric neurologist, is evaluated by the researcher. A second evaluation is repeated one week later after a follow-up examination to ensure test-retest reliability.
  The Hypertonia Assessment Tool (HAT) was developed to address the need for a single instrument capable of evaluating different subtypes of increased muscle tone within one assessment battery. The HAT involves observing a patient's limb during a targeted passive stretch and during voluntary movement to assess increased tone or resistance. The scale consists of seven items in total: two assess spasticity, two assess rigidity, and three assess dystonia.

CONTACTS AND LOCATIONS:
Overall Officials: Bulent Elbasan, Prof. Dr., Study Chair — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
All IPD collected throughout the trial, only IPD used in the results publication.

REFERENCES:
- [Result] Marsico P, Frontzek-Weps V, Balzer J, van Hedel HJ. Hypertonia Assessment Tool. J Child Neurol. 2017 Jan;32(1):132-138. doi: 10.1177/0883073816671681. Epub 2016 Oct 15. PMID 27742862
- [Result] Jethwa A, Mink J, Macarthur C, Knights S, Fehlings T, Fehlings D. Development of the Hypertonia Assessment Tool (HAT): a discriminative tool for hypertonia in children. Dev Med Child Neurol. 2010 May;52(5):e83-7. doi: 10.1111/j.1469-8749.2009.03483.x. PMID 20540176
- [Result] Haberfehlner H, Goudriaan M, Bonouvrie LA, Jansma EP, Harlaar J, Vermeulen RJ, van der Krogt MM, Buizer AI. Instrumented assessment of motor function in dyskinetic cerebral palsy: a systematic review. J Neuroeng Rehabil. 2020 Mar 5;17(1):39. doi: 10.1186/s12984-020-00658-6. PMID 32138731
- [Result] Hadders-Algra M. Early Diagnostics and Early Intervention in Neurodevelopmental Disorders-Age-Dependent Challenges and Opportunities. J Clin Med. 2021 Feb 19;10(4):861. doi: 10.3390/jcm10040861. PMID 33669727